CLINICAL TRIAL: NCT00810316
Title: Evaluate The Pharmacokinetics Of Two Alprazolam Formulations (Immediate Release And Extended Release Tablets) And A Clonazepam Tablet In A Healthy Mexican Population
Brief Title: Evaluate Pharmacokinetics Of Two Different Pharmaceutical Oral Formulations Of Alprazolam And A Clonazepam Tablet In Mexican Healthy Population
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: A6131015
Record Dates: First submitted 2008-12-16; First posted 2008-12-18 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Pharmacokinetics
Keywords: Alprazolam; Alprazolam extended release; Clonazepam; Pharmacokinetics; Mexican population; Healthy
MeSH Terms: interventions — Alprazolam; Clonazepam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Other)
  Interventions: Drug: Alprazolam
- Treatment B (Other)
  Interventions: Drug: Alprazolam XR
- Treatment C (Other)
  Interventions: Drug: Clonazepam

INTERVENTIONS:
Drug: Alprazolam — Administration of a single oral dose tablet of 1 mg of alprazolam immediate release on Day 1 morning, between 8-9 am with 250 ml of water in at least 10 hours of fasting conditions
  Other Names: Tafil, Xanax
  Arms: Treatment A
Drug: Alprazolam XR — Administration of a single oral dose tablet of 1 mg of alprazolam modified release on Day 1 morning, between 8-9 am with 250 ml of water in at least 10 hours of fasting conditions
  Other Names: Tafil AP, Xanax XR
  Arms: Treatment B
Drug: Clonazepam — Administration of a single oral dose of two tablets of 0.5 mg of clonazepam on Day 1 morning, between 8-9 am with 250 ml of water in at least 10 hours of fasting conditions
  Other Names: Rivotril
  Arms: Treatment C

SUMMARY:
To estimate the pharmacokinetics of single doses of benzodiazepines in Mexican adult healthy volunteers: a) alprazolam tablet extended release, b) alprazolam tablet immediate release, and clonazepam tablet.

DETAILED DESCRIPTION:
To determine pharmacokinetics of alprazolam and clonazepam in Latin-American population; in Mexico, both drugs are still widely used as first or second choice in the treatment of anxiety disorders.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteers aged between 18 and 40 years old.

Exclusion Criteria:

* Subjects presenting changes on their vital signs constants registered at volunteers' screening.
* Volunteers with any of the following: noncompliance of proposed inclusion criteria; requiring another drug product throughout the study conduction; pregnant or nursing females; history of cardiovascular, renal, hepatic, muscular, metabolic, gastrointestinal, neurological, endocrine, psychiatric, hematopoietic or any other anemia kind, disease, asthma, or organic disorder; history of dyspepsia, gastritis, esophagitis, duodenal or gastric ulcer or any condition possibly affecting drug absorption; history of acute narrow or glaucoma; exposed to drug products known as hepatic enzyme or inductors; who had received any drug product within 14 days or 5 half lives; who had been hospitalized due to any problem within 60 days prior to study start; history of sensitivity to BZD; who had drink alcohol or any beverage containing xanthines or who had taken smoked food or grapefruit juice within 72 hours prior to start hospitalization period, who had blood donated or lost 450 mL or more within 60 days prior to study start; requiring any special diet regardless the cause.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
AUC last: Area under the curve of plasma concentration from administration up to time t (last sampling timepoint) calculated by trapezoid method. | Sampling times: 0 to 96 hours
AUC inf: Area under the curve of plasma concentration from administration up to infinitum extrapolated time. | Sampling times: 0 to 96 hours
Cmax: Maximum plasma concentration graphically obtained, based on plasma concentration versus time profile. | Sampling times: 0 to 96 hours
t 1/2: Half life time. | Sampling times: 0 to 96 hours
Tmax: Time from administration up to maximum plasma concentration, graphically obtained based on plasma concentration versus time profile. | Sampling times: 0 to 96 hours

SECONDARY OUTCOMES:
No Secondary Outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Col. Arenal Tepepan, Mexico City, Mexico

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6131015&StudyName=Evaluate%20Pharmacokinetics%20Of%20Two%20Different%20Pharmaceutical%20Oral%20Formulations%20Of%20Alprazolam%20And%20A%20Clonazepam%20Tablet%20In%20Mexican%20Healthy%20Populat